CLINICAL TRIAL: NCT03449095
Title: Examining the Impact of Stress on the Emotionally Reinforcing Properties of Alcohol in Heavy Social Drinkers: A Multimodal Investigation Integrating Laboratory and Ambulatory Methods
Brief Title: Understanding Alcohol Reward in Social Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Catharine Fairbairn, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: R01AA025969 (NIH)
Record Dates: First submitted 2017-11-23; First posted 2018-02-28 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder; Alcohol Intoxication; Alcohol; Harmful Use; Alcoholism; Binge Drinking
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Alcoholic Intoxication; Binge Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Administration (Experimental): A moderate dose of alcohol (Target BAC .08%)
  Interventions: Drug: Alcohol
- Control Beverage Administration (No Intervention): Participants consume a non-alcoholic beverage

INTERVENTIONS:
Drug: Alcohol — Alcohol Target BAC .08%
  Arms: Alcohol Administration

SUMMARY:
In this study, the investigators examine whether emotional and social reward from alcohol varies depending on the social context of consumption.

DETAILED DESCRIPTION:
Objective: Although the vast majority of alcohol consumption outside the laboratory occurs in social context, experimental studies of alcohol's emotionally reinforcing effects have overwhelmingly examined individuals drinking in isolation. The current study examines motivationally salient elements of everyday social drinking contexts as moderators of alcohol-related reinforcement. More specifically, the present study examine whether alcohol is more reinforcing within the context of unfamiliar vs. familiar social interaction and, further, whether alcohol is more reinforcing within the context of low vs. high quality social relationships. The current study furthermore examine whether individuals with characteristics that put them at risk for developing an alcohol use disorder (e.g., male gender, impulsive/extraverted personality profile, heavy patterns of consumption, family history of AUD, ...) exhibit heightened emotional reinforcement from alcohol within these social drinking contexts.

The current project represents a test of competing theories of alcohol reinforcement. Alcohol myopia theory-which has heretofore represented the most prominent theory of alcohol's effects-predicts that alcohol's ability to relieve stress depends on the nature (positive or negative) of stimuli in the drinker's immediate environment. Alcohol myopia theory might thus predict that alcohol's rewarding effects will be larger within familiar interactions and within secure relationships. In contrast, the social attributional theory of alcohol reinforcement predicts that alcohol-related reinforcement will be most pronounced within the context of unfamiliar social interactions.

In addition to providing an opportunity to test contextual and individual-level moderators of alcohol reinforcement, the current study represents an opportunity to directly test the replicability of research indicating a pronounced reinforcing effect of alcohol specifically within interactions among unfamiliar individuals (Sayette et al., 2012; Fairbairn et al., 2013).

Study Population: Participants will consist of 640 male and female drinkers, aged 21-30, with no reported history of severe alcohol use disorder. Participants will be sampled such that at least 360 of these participants will classify as heavy drinkers.

Design: In the laboratory arm of the study, individuals will be randomly assigned to consume either a moderate dose of alcohol or a control beverage in the company of either familiar or unfamiliar individuals. Of these individuals, a subset will participate in additional tasks post beverage-consumption including a hyperscanning EEG task, while an additional subset will also participate in an ambulatory assessment period over the course of several weeks to examine the interaction of alcohol and social contextual factors in daily life. In the ambulatory study arm, participants will wear transdermal sensors to assess BAC and will further provide information about their mood and their social contexts in response to random prompts.

Outcome Measures: Primary outcome measures include self-reports of positive and negative mood and perceived social reinforcement. The investigators will also examine facial expressions using the Facial Action Coding System, a comprehensive, anatomically-based system for categorizing facial muscle movement. One aim of the current study is to examine whether differential reinforcement from alcohol in unfamiliar social contexts emerges only with respect to self-reports, or is also observable within facial behaviors. EEG/ERP measures will also be examined for a subset of participants engaged in a hyperscanning task.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21 and 30
* Currently drinks alcohol
* Able to provide at least 2 same-gender friend referrals

Exclusion Criteria:

* Female participant is pregnant or trying to become pregnant
* Endorsed medical disorder caused by, or made worse by, alcohol
* History of severe alcohol problems
* Use of drugs known to interact with alcohol

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — May be either male or female, but must be same as gender assigned at birth.
Enrollment: 640 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catharine E Fairbairn, Ph.D., Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Champaign, Illinois, United States

REFERENCES:
- [Background] Steele CM, Josephs RA. Alcohol myopia. Its prized and dangerous effects. Am Psychol. 1990 Aug;45(8):921-33. doi: 10.1037//0003-066x.45.8.921. PMID 2221564
- [Background] Fairbairn CE. Drinking among strangers: A meta-analysis examining familiarity as a moderator of alcohol's rewarding effects. Psychol Addict Behav. 2017 May;31(3):255-264. doi: 10.1037/adb0000264. Epub 2017 Mar 13. PMID 28287750
- [Background] Fairbairn CE, Sayette MA. A social-attributional analysis of alcohol response. Psychol Bull. 2014 Sep;140(5):1361-82. doi: 10.1037/a0037563. PMID 25180806
- [Background] Sayette MA, Creswell KG, Dimoff JD, Fairbairn CE, Cohn JF, Heckman BW, Kirchner TR, Levine JM, Moreland RL. Alcohol and group formation: a multimodal investigation of the effects of alcohol on emotion and social bonding. Psychol Sci. 2012 Aug 1;23(8):869-78. doi: 10.1177/0956797611435134. Epub 2012 Jul 3. PMID 22760882
- [Background] Fairbairn CE, Sayette MA. The effect of alcohol on emotional inertia: a test of alcohol myopia. J Abnorm Psychol. 2013 Aug;122(3):770-81. doi: 10.1037/a0032980. PMID 24016015

RESULTS

PARTICIPANT FLOW:
Groups:
- Alcohol Administration: Primary participants in the current study consisted of both eligible individuals who first contacted the lab and their eligible friends. Here we report the total number of individual participants (both initial contacts and their friends) who received a moderate dose of alcohol (Target BAC .08%).
- Control Beverage Administration: Primary participants in the current study consisted of both eligible individuals who first contacted the lab and their eligible friends. Here we report the total number of individual participants (both initial contacts and their friends) who received a non-alcoholic beverage.
Period: Overall Study
Arm/Group | Alcohol Administration | Control Beverage Administration
Started | 320 | 320
Completed | 320 | 320
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Primary participants in the current study consisted of both eligible individuals who first contacted the lab and their eligible friends. Here we report the total number of individual participants (both initial contacts and their friends) enrolled in the study.
Groups:
- Alcohol Administration: Primary participants in the current study consisted of both eligible individuals who first contacted the lab and their eligible friends. Here we report the data from individual participants (both initial contacts and their friends) who received a moderate dose of alcohol (Target BAC .08%).
- Control Beverage Administration: Primary participants in the current study consisted of both eligible individuals who first contacted the lab and their eligible friends. Here we report the data from individual participants (both initial contacts and their friends) who received a non-alcoholic beverage.
- Total: Total of all reporting groups
Arm/Group | Alcohol Administration | Control Beverage Administration | Total
Number analyzed (Participants) | 320 | 320 | 640
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.63 (1.923) | 22.74 (2.101) | 22.69 (2.013)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 160 | 320
  Male | 160 | 160 | 320
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66 | 68 | 134
  Not Hispanic or Latino | 254 | 252 | 506
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 110 | 129 | 239
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 180 | 164 | 344
  More than one race | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 320 | 320 | 640
Education level [Mean (Standard Deviation); unit: Years of Education] | 16.08 (1.716) | 16.09 (1.741) | 16.08 (1.727)

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Emotion
Description: Positive and negative emotion will be assessed during the laboratory beverage-administration session via self-report on the "8-item Mood Measure." This measure yields two subscales (positive emotion; negative emotion) each ranges from 1 to 6. For positive mood, higher value represents increased alcohol reward. For negative mood, lower value represents increased alcohol reward.
Time Frame: during the laboratory session, up to 9 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alcohol Administration | Control Beverage Administration
Number analyzed (Participants) | 320 | 320
score on a scale
  Positive Emotion | 3.49 (1.085) | 2.98 (1.101)
  Negative Emotion | 0.32 (0.447) | 0.673 (0.750)
Statistical Analysis 1: Comparison: Alcohol Administration vs Control Beverage Administration; Test type: Superiority; p < 0.001, ANOVA — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance

2. Primary Outcome: Self-Reported Social Reinforcement
Description: Social reinforcement will be assessed using an index of perceived social closeness as well as a modified version of the Perceived Group Reinforcement Scale. The score of the scale ranges from 1 to 9. Higher score indicates increased alcohol reward.
Time Frame: during the laboratory session, up to 9 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alcohol Administration | Control Beverage Administration
Number analyzed (Participants) | 320 | 320
score on a scale | 7.471 (1.129) | 7.180 (1.155)
Statistical Analysis 1: Comparison: Alcohol Administration vs Control Beverage Administration; Test type: Superiority; p = .001, ANCOVA — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance

3. Secondary Outcome: Social Bonding
Description: Social bonding will be assessed during the laboratory beverage-administration session. This will be assessed by examining the synchronization among group members of facial expressions of emotion.
Time Frame: 1 day (laboratory session)
Reporting Status: Not Posted

4. Secondary Outcome: Self-Reported Emotion
Description: Positive and negative emotion will be assessed during the ambulatory assessment period via self-report on the "8-item Mood Measure."
Time Frame: 2-3 week ambulatory assessment period
Reporting Status: Not Posted

5. Secondary Outcome: Interpersonal Distance
Description: Physical proximity to other participants during the experiment
Time Frame: 1 day (laboratory session)
Reporting Status: Not Posted

6. Secondary Outcome: Neuro-cognitive Social Engagement
Description: Electroencephalogram (EEG) hyperscanning methods will be employed to assess task engagement and social attention, including through the examination of event-related potentials (ERPs) during social tasks.
Time Frame: 1 day (laboratory session)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6-9 hours (length of the laboratory session)
Description: The intervention of the study is laboratory alcohol administration.
Groups:
- Alcohol Administration: Primary participants in the current study consisted of both eligible individuals who first contacted the lab and their eligible friends. Here we report the number of individual participants (both initial contacts and their friends) who received a moderate dose of alcohol (Target BAC .08%).
- Control Beverage Administration: Primary participants in the current study consisted of both eligible individuals who first contacted the lab and their eligible friends. Here we report the number of individual participants (both initial contacts and their friends) who received a non-alcoholic beverage.
Arm/Group | Alcohol Administration | Control Beverage Administration
All-Cause Mortality (participants affected / at risk) | 0/320 | 0/320
Serious Adverse Events (participants affected / at risk) | 0/320 | 0/320
Other Adverse Events (participants affected / at risk) | 0/320 | 0/320

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT03449095/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03449095/ICF_000.pdf